CLINICAL TRIAL: NCT07029880
Title: Clinical Performance of Metal Ceramic Fixed Dental Prostheses Using Two Porcelain Veneering Systems: A Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Inas Adel Mahmoud, The principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01008402645
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Teeth Requiring Fixed Metal Ceramic Prosthesis
MeSH Terms: interventions — Resin Cements

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metal ceramic fixed dental prosthesis veneered using Vintage Pro and cemented with BeautiLink SA cem (Experimental): full veneered metal ceramic dental prosthesis cemented with resin cement
  Interventions: Other: full veneered metal ceramic dental prosthesis cemented with resin cement
- metal ceramic fixed dental prosthesis veneered using IPS style ceram and cemented with BeautiLink SA (Active Comparator): full veneered metal ceramic dental prosthesis cemented with resin cement
  Interventions: Other: full veneered metal ceramic dental prosthesis cemented with resin cement

INTERVENTIONS:
Other: full veneered metal ceramic dental prosthesis cemented with resin cement — full veneered metal ceramic dental prosthesis cemented with resin cement

SUMMARY:
This study aims to evaluate the clinical performance of metal ceramic fixed dental prostheses veneered with two porcelain systems; Vintage Pro and IPS style ceram and cemented with Beautilink SA cement.

ELIGIBILITY:
1. Age ≥ 21 years
2. Vital or endodontically treated teeth
3. Abutments with no mobility
4. Abutments with adequate crown/root ratio more than 1:1
5. Willing and able to provide written informed consent
6. Ability to attend all follow-up appointments
7. Adequate oral hygiene as determined by the investigator

And the following exclusion criteria:

1. Patients with active periodontal disease (probing depth > 4mm, bleeding on probing)
2. Patients with parafunctional habits (e.g., bruxism confirmed by clinical examination)
3. Poor oral hygiene (plaque index > 30%)
4. Pregnancy or nursing
5. Systemic diseases affecting treatment outcomes (e.g., uncontrolled diabetes, immunosuppression)
6. Known allergies to study materials (alloy, ceramic, or resin cement components)
7. Inability to comply with study requirements
8. Current participation in other dental clinical trials
9. Active orthodontic treatment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Wear | 18 months
  Measuring device :Digital software (Geomagic) .Measuring Unit :Root mean square

SECONDARY OUTCOMES:
Restoration Failure | 18 months
  Measuring device: Modified USPHS criteria.Measuring Unit:Alpha: none Bravo: Discrete crack .Charlie: Chipping.Delta: Bulk fracture
Luster of restoration | 18 months
  Measuring device:Modified USPHS criteria Measuring Unit :Alpha: restoration is shiny has enamel like translucent surface.Bravo: restoration is dull and somewhat opaque .Charlie: restoration surface is distinctly dull and opaque.
Color match | 18 months
  Measuring device:Modified USPHS criteria. Measuring Unit:Alfa: no mismatch in color, shade and translucency between restoration and adjacent teeth Bravo: slight mismatch.Charlie: esthetically unacceptable mismatch
Surface texture | 18 months
  Measuring device:Modified USPHS criteria.Measuring Unit:Alfa: Smooth, glazed or glossy surface.Bravo: Slightly rough surface.Charlie: Very rough surface

CONTACTS AND LOCATIONS:
Overall Officials: faculty of dentisry cairo university, Principal Investigator — Cairo University; faculty of dentisry cairo university, Principal Investigator — unaffliated
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided